CLINICAL TRIAL: NCT00939445
Title: Short Daily Hemodialysis and Online HDF: Which One is Better?
Acronym: SHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VJR-NEPHRO001
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online HDF (Active Comparator): Online HDF
  Interventions: Procedure: Online HDF
- Short Daily Hemodialysis (Active Comparator): Short Daily Hemodialysis
  Interventions: Procedure: Short Daily Hemodialysis

INTERVENTIONS:
Procedure: Online HDF — Online HDF
  Arms: Online HDF
Procedure: Short Daily Hemodialysis — Short Daily Hemodialysis
  Arms: Short Daily Hemodialysis

SUMMARY:
1. To compare the efficacy of

1. Short Daily Hemodialysis
2. Online HDF in term of adequacy of dialysis.

DETAILED DESCRIPTION:
The investigators intend to compare the efficacy between these modalities of treatment in terms of adequacy and also other parameters such as calcium-phosphorus balance and hematocrit

ELIGIBILITY:
Inclusion Criteria:

* stable ESRD
* KT/V > 1.2 for thrice weekly or > 1.8 for twice weekly

Exclusion Criteria:

* Inadequate vascular access flow rate
* Concurrent medical illnesses
* History of non-compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Adequacy | 3 months

SECONDARY OUTCOMES:
Hematocrit, calcium, phosphorus | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Unit, BMA Medical College and Vajira Hospital, Bangkok, Thailand